CLINICAL TRIAL: NCT05997017
Title: A Phase 2 Multi-center Open-label Trial of Nab-Sirolimus in Combination With Letrozole in Advanced or Recurrent Endometrioid Endometrial Cancer
Brief Title: Trial of Nab-Sirolimus in Combination With Letrozole in Patients With Advanced or Recurrent Endometrioid Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EEC-201
Record Dates: First submitted 2023-08-10; First posted 2023-08-18 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Cancer; Endometrioid Tumor; Cancer; Tumor; Recurrent Endometrial Carcinoma; Endometrioid Endometrial Cancer
Keywords: nab-Sirolimus; FYARRO; Letrozole; Endometrial; Recurrent; ABI-009; Endometrial Carcinoma; Endometrioid Tumor; Endometrial Cancer; Recurrent Endometrial Carcinoma; Endometrioid Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endometrioid Endometrial Cancer (Experimental): Patients with advanced or recurrent endometrioid endometrial carcinoma
  Interventions: Drug: nab-sirolimus

INTERVENTIONS:
Drug: nab-sirolimus — Prospective Phase 2, open-label, multi-institutional study to evaluate the efficacy and safety of nab-sirolimus + letrozole in patients
  Other Names: ABI-009

SUMMARY:
A Phase 2 Multi-center Open-label Trial of nab-Sirolimus in Combination with Letrozole in Advanced or Recurrent Endometrioid Endometrial Cancer

DETAILED DESCRIPTION:
This is a prospective phase 2, open-label, multi-institutional study to evaluate the efficacy and safety of nab-sirolimus + letrozole in patients with advanced or recurrent endometrioid endometrial carcinoma who have received 0-1 prior lines of chemotherapy in the recurrent/metastatic setting. Patients will be treated with nab-sirolimus (given IV on Days 1 and 8 in a 21-day cycle, combined with letrozole (orally, daily) until unacceptable toxicity or disease progression, or until in the opinion of the Investigator the patient is no longer benefiting from therapy, or at patient discretion.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have clinically confirmed advanced or recurrent endometrioid endometrial carcinoma. Histologic documentation of the recurrence is suggested but not required.
2. All patients must have 1 or more measurable target lesion at baseline by computed tomography (CT; or magnetic resonance imaging [MRI] if CT scans are contraindicated) as defined by RECIST version 1.1.
3. Patients must have EEC that is metastatic or locally advanced where surgical resection is not an option or likely to result in severe morbidity.
4. Prior treatment history:

   1. Adjuvant setting - treatment with chemotherapy, hormonal therapy,checkpoint inhibitors, and/or other therapy is permitted as long as theadjuvant therapy ended ≥6 months from enrollment.
   2. Recurrent/advanced/metastatic setting - treatment with 0-1 prior chemotherapy regimens is permitted (patients may be naïve to chemotherapy); chemotherapy must have been completed ≥3 months prior to enrollment. Patients are permitted to have received adjuvant chemotherapy and no more than 1 line of chemotherapy in the recurrent/advanced/metastatic setting.
   3. Non-chemotherapy-based treatment (eg, checkpoint inhibitors, hormonal therapy, and/or small molecule agents) is permitted at any point as long as therapy ended ≥4 weeks prior to enrollment.
   4. Patients who have received prior therapy in the recurrent/advanced/metastatic setting must have achieved a complete or partial response(investigator-assessed) to at least 1 therapy.
5. Age: 18 years or older.
6. Patient must have Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
7. Adequate liver function:

   1. Total bilirubin ≤1.5 × upper limit of normal (ULN) (unless due to Gilbert's syndrome, then ≤3 × ULN)
   2. Aspartate aminotransferase (AST) ≤2.5 × ULN (≤5 × ULN if attributable to liver metastases)
8. Adequate renal function: creatinine clearance (CrCL) ≥30 mL/min based on Cockcroft-Gault
9. Adequate hematologic parameters:

   1. Absolute neutrophil count (ANC) ≥1.0 × 109/L (growth factor support allowed)
   2. Platelet count ≥100,000/mm3 (100 × 109/L) (transfusion and/or growth factor support allowed)
   3. Hemoglobin ≥8.0 g/dL (transfusion and/or growth factor support allowed)
10. Fasting serum triglyceride must be ≤300 mg/dL; fasting serum cholesterol must be less than or equal to 350 mg/dL.
11. Minimum of 4 weeks since any major surgery, completion of radiation, or completion of prior systemic anticancer therapy, or at least 5 half-lives if the prior therapy is a single agent small-molecule therapeutic, and adequately recovered from the acute toxicities of any prior therapy, including neuropathy, to Grade ≤1.
12. Non-pregnant and non-breastfeeding female:

    1. Females of childbearing potential must agree to use effective contraception or abstinence without interruption from 28 days prior to starting nab-Sirolimus through 3 months after the last dose of nab-Sirolimus and have a negative serum pregnancy test (beta human chorionic gonadotropin [β-hCG]) result at screening and agree to ongoing pregnancy testing during the course of the study, and after the end of study treatment. A second form of birth control is required even if she has had a tubal ligation.
    2. Sexual abstinence is considered a highly effective contraceptive method only if defined as refraining from heterosexual intercourse from 28 days prior to starting study medication throughout 3 months after last dose of study medication. The reliability of sexual abstinence should be evaluated in relation to the duration of the study and the preferred and usual lifestyle of the patient.
13. The patient understands and signs the informed consent.
14. Willingness and ability to comply with scheduled visits, laboratory tests, and other study procedures.
15. Patients with a known history of human immunodeficiency virus (HIV)infection are eligible if:

    1. There has been no acquired immunodeficiency syndrome (AIDS)-defining opportunistic infection in 12 months prior to enrollment.
    2. The patient has been receiving an antiretroviral therapy regimen for≥4 weeks and the HIV viral load is <400 copies/mL prior to enrollment.
    3. Antiretroviral therapy regimen does not include strong cytochrome(CYP)3A4 inhibitors or inducers

Exclusion Criteria:

1. Prior treatment with an mTOR inhibitor, including nab-sirolimus.
2. Patients with known inactivating TSC1 or TSC2 alterations (based on tissue or liquid next generation sequencing [NGS]) unless the PRECISION 1 study (NCT05103358) has been closed to enrollment.
3. Severe (Grade ≥3) ongoing infection requiring parenteral or oral anti-infective treatment, either ongoing or completed ≤7 days prior to enrollment.
4. Patients with primary refractory disease (ie, those who have never achieved a complete or partial response to prior therapy) are not permitted on study.
5. Patients with the following are excluded:

   1. Known or suspected brain metastases.
   2. Severe heart disease defined as unstable angina pectoris, New York Heart Association (NYHA) Class III or IV congestive heart failure, myocardial infarction ≤6 months prior to first study treatment, serious uncontrolled cardiac arrhythmia or any other clinically significant cardiac disease.
   3. Severe lung disease defined as a diffusing capacity for carbon monoxide (DLCO) that is ≤50% of normal predicted value and/or an O2 saturation ≤88% at rest on room air (Note: spirometry and pulmonary function tests [PFTs] are not required to be performed unless clinically indicated).
   4. Nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the treatment with the study therapy.
   5. A history of malignancies other than the one under treatment unless the patient is disease-free for more than 5 years from completion of therapy administered with curative intent. Controlled non-melanoma skin cancers, carcinoma in situ of the cervix, resected incidental prostate cancer, certain low grade hematologic malignancies (eg, chronic lymphocytic leukemia [CLL], follicular lymphoma, etc), or other adequately treated carcinoma in situ may be eligible, after discussion with the Medical Monitor.
   6. Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg
   7. Patients with history of interstitial lung disease and/or pneumonitis, or pulmonary hypertension.
   8. Active hepatitis B and/or hepatitis C infection and detectable viral load despite antiviral therapy
6. Required use of concomitant medications with strong CYP3A4 interactions (induction or inhibition) should be discontinued (strong inhibitors include ketoconazole, itraconazole, voriconazole, erythromycin, clarithromycin, telithromycin; strong inducers include rifampin and rifabutin). These agents must be discontinued prior to first dose of nab-sirolimus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 29 (Estimated)
Dates: Start 2023-12-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 12 Months
  ORR, defined as the proportion of patients with best overall response (BOR) of confirmed partial response (PR) or complete response (CR) from the time of study treatment initiation until progression of disease (PD) as determined by the Investigator using RECIST v1.1.

SECONDARY OUTCOMES:
Duration of response (DOR) | 12 Months
  Determined for patients with BOR of confirmed CR or PR
Disease Control Rate (DCR): CR or PR | 12 Months
  BOR of confirmed CR or PR (either of any duration) or stable disease (SD) following study treatment initiation (by IRR)
Time to response (TTR) | 12 Months
  Time from study treatment initiation to initial measurement of CR or PR, where CR or PR is subsequently confirmed
Progression-free survival (PFS) | 12 Months
  Number of months from study treatment initiation to the date of disease progression 3 or death due to any cause
Overall survival (OS) | 24 Months
  Number of months from study treatment initiation to the date of death due to any cause or last follow up date if alive
Incidence and severity | 12 Months
  Of treatment-emergent and treatment-related adverse events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Willis Navarro, MD, Study Director — Aadi Bioscience
Locations (9):
- United States (9):
  - Michael Birrer, MD, PhD, Little Rock, Arkansas
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Oklahoma University Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Women & Infants Hospital, Providence, Rhode Island
  - Texas Oncology - Tyler, Tyler, Texas
  - Swedish Cancer Institute, Seattle, Washington